CLINICAL TRIAL: NCT07357506
Title: Mitigating Cutaneous Toxicity in Patients Undergoing TomoTherapy; A Randomized Controlled Trial of Skin-Protective Strategies
Brief Title: Reducing Skin Side Effects in Patients Receiving Radiation on Tomotherapy
Acronym: MCTPUT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Zaheeda Mulla, Supervisor, King Faisal Specialist Hospital & Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RAC#: 2251649
Record Dates: First submitted 2025-11-26; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Radiotherapy; Dermatitis
MeSH Terms: conditions — Head and Neck Neoplasms; Dermatitis

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in parallel groups to receive either Mepitel or a fragrance-free emollient as a skin-protective strategy during TomoTherapy. Each participant will receive only one of the two interventions throughout the study period, and outcomes will be compared between groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: STDoC + fragrance-free emollient (glycerol-based) from day 1 + absorbent polyurethane foam dr (Active Comparator): Participants in Arm A will receive standard treatment during TomoTherapy (STDoC) plus a fragrance-free, glycerol-based emollient applied to skin starting day 1 of treatment. If participants develop Grade ≥2 radiation dermatitis, an absorbent polyurethane foam dressing (PolyMem-equivalent) will be applied to the affected area. This arm serves as the active comparator for evaluating the efficacy of the experimental intervention (Mepitel).
  Interventions: Other: Fragrance-Free Emollient (Glycerol-Based); A fragrance-free, glycerol-based emollient applied to the skin from day 1 of TomoTherapy.
- Arm B: STDoC + silicone-based semi-permeable barrier film (Mepitel Film-equivalent) applied from day (Experimental): A silicone-based semi-permeable barrier film applied to the skin from day 1 of TomoTherapy. Evaluated as the experimental intervention to prevent or reduce radiation-induced skin toxicity.
  Interventions: Device: Mepitel Film (Silicone-Based Semi-Permeable Barrier Film)

INTERVENTIONS:
Other: Fragrance-Free Emollient (Glycerol-Based); A fragrance-free, glycerol-based emollient applied to the skin from day 1 of TomoTherapy. — A foam dressing applied to areas of Grade ≥2 radiation dermatitis for skin protection during TomoTherapy. Part of Arm A.
  Arms: Arm A: STDoC + fragrance-free emollient (glycerol-based) from day 1 + absorbent polyurethane foam dr
Device: Mepitel Film (Silicone-Based Semi-Permeable Barrier Film) — A silicone-based semi-permeable barrier film applied to the skin from day 1 of TomoTherapy. Evaluated as the experimental intervention to prevent or reduce radiation-induced skin toxicity.
  Arms: Arm B: STDoC + silicone-based semi-permeable barrier film (Mepitel Film-equivalent) applied from day

SUMMARY:
* Radiation dermatitis is a common side effect in head and neck cancer (HNC) patients receiving radiotherapy, especially with advanced techniques like TomoTherapy. The use of 6 MegaVoltage (MV) Flattening Filter-Free (FFF) beams and shorter Source to Skin Distance (SSD) in TomoTherapy may increase skin dose, leading to higher rates of skin reactions such as redness, irritation, and pain. These reactions can affect patient comfort, increase the risk of infection, and even interrupt treatment.
* Although radiation dermatitis is frequent, there is no widely accepted standard for preventing or managing it. Supportive care programs, like the Dermatitis Control Program (DeCoP), and other supportive care programs using silicone-based semi-permeable barrier film have shown that simple measures-such as good skin hygiene and keeping the skin moist, can help reduce skin damage during treatment.
* This study will evaluate the effectiveness of fragrance-free emollient (glycerol-based) + absorbent polyurethane foam dressing versus silicone-based semi-permeable barrier film dressing in preventing or reducing skin toxicity in HNC patients receiving TomoTherapy. These products are easy to apply, affordable, and widely available, making them practical options for routine care.

DETAILED DESCRIPTION:
Background/Introduction; Head and neck cancers (HNC) are frequently treated with definitive radiotherapy or chemoradiotherapy, which are effective modalities for tumor control and organ preservation. However, these treatments are often associated with significant acute toxicities, particularly incidence of radiation dermatitis which is as high as 84%. Radiation-induced skin reactions are typically classified as acute, consequential-late, or chronic, with acute dermatitis being the most immediate and impactful during treatment. Studies reveal that acute radiation-dermatitis (ARD) occur within 24 hours but usually begin within days to weeks of initiating radiotherapy and is responsible for discomfort, pain, aesthetic changes, increased risk of infection, and potentially, treatment interruptions, thereby affecting both the patient's quality of life and therapeutic outcomes.

* Despite the clinical burden of radiation dermatitis, there is currently no universally accepted standard for its prevention or management. Established evidence supports the effectiveness of simplified, supportive care approaches, such as the Dermatitis Control Program (DeCoP), which focus on basic skin hygiene and maintaining a moist wound-healing environment during radiotherapy. This program demonstrated favorable outcomes in managing radiation dermatitis in patients with head and neck cancer.
* Clinical studies demonstrated that Moisturized skin care effectively reduced the severity and delayed the onset of radiation dermatitis, while also slowing down the decrease in skin moisture during radiotherapy.
* Additionally, barrier films such as Mepitel Film have shown promise in reducing ARD severity and moist desquamation. Systematic reviews and feasibility trials report benefit in breast and head/neck cancer patients. Including Mepitel Film as a comparator allows direct head-to-head testing of two evidence-based, guideline-consistent strategies.
* TomoTherapy, is a highly conformal and image-guided intensity-modulated radiotherapy (IMRT) technique. The system has shorter Source to Skin Distance (SSD) of 85cm and uses 6 MegaVoltage (MV) Flattening Filter-Free (FFF) energy which will increase the low energy photon contribution. Subsequently, one of the common side effects associated with this treatment is cutaneous toxicity, which can lead to skin irritation, erythema, and ulceration.

Hypothesis

* Use of fragrance-free emollient with absorbent dressing OR silicone barrier film, will reduce the severity of acute radiation dermatitis (ARD) with differential effects between interventions.
* While ARD significantly impacts patient well-being and clinical outcomes, standardized preventive care protocols remain inconsistent or under-researched in TomoTherapy. This study addresses that gap by evaluating a practical, low-cost intervention- fragrance-free emollient (glycerol-based) from day 1 + absorbent polyurethane foam dressing versus silicone-based semi-permeable barrier film applied from day 1-for its effectiveness in reducing skin toxicity and improving patient quality of life during TomoTherapy.

Methodology This is a prospective, randomized, controlled, two-arm clinical trial evaluating strategies to mitigate radiation-induced skin toxicity in head and neck cancer (HNC) patients undergoing TomoTherapy.

Design:

Parallel-group design with 1:1 allocation using computer-generated block randomization, stratified by chemotherapy status.

Masking:

Open-label design; outcome assessors (radiation oncologists grading dermatitis) will be blinded where feasible.

Sample Size:

Approximately 104 patients (52 per arm) to detect a 20% absolute reduction in Grade ≥2 dermatitis incidence (from 55% to 35%) with 80% power and α = 0.05, accounting for 10% attrition.

Data Collection:

Weekly (Day 1,7,14,21,28,35) CTCAE skin assessments documented in MOSAIQ. QoL instruments (EORTC QLQ-C30 v3 and QLQ-HN35) administered at Baseline (Day 1), mid-treatment (Day 17), and end-of-treatment (Day 35).

Clinical and treatment data recorded in an encrypted Excel database.

Ethical Considerations:

All participants receive at least standard of care (STDoC). Written informed consent required prior to radiotherapy. Data are anonymized and securely stored.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 80 with newly diagnosed head and neck (H&N) carcinoma (confirmed by pathology)
* Must be receiving radiotherapy using Tomotherapy

Exclusion Criteria:

* Prior H&N radiotherapy
* pre-existing skin disease
* allergy to study products.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients developing Common Terminology Criteria for Adverse Events (CTCAE) v5.0 Grade ≥2 dermatitis by completion of radiotherapy. | Day 7,14,21,28,35 of radiotherapy for all patients registered in the study
  Clinical evaluation of radiation-induced dermatitis will be measured using the Common Terminology Criteria for Adverse Events (CTCAE) version [v5.0], focusing specifically on radiation dermatitis grading (21).
  * Radiation dermatitis will be assessed weekly (Day 7,14,21,28,35) by the attending radiation oncologist throughout the course of treatment, with documentation in MOSAIQ (radiation oncology information system) of onset, peak severity, and any treatment-related complications or interruptions.
  * CTCAE grading will be used to classify skin reactions as follows:
  * Grade 1: Faint erythema or dry desquamation
  * Grade 2: Moderate to brisk erythema; patchy moist desquamation mostly in skin folds
  * Grade 3: Moist desquamation in non-skin-fold areas; bleeding with minor trauma
  * Grade 4: Skin necrosis or ulceration of full-thickness dermis
  * Grade 5: Death (extremely rare in this context)

SECONDARY OUTCOMES:
-Number of days to start of Grade ≥2 dermatitis between arms. | Day 7,14,21,28,35 during the course of radiotherapy
  Clinical evaluation of radiation-induced dermatitis will be measured using the Common Terminology Criteria for Adverse Events (CTCAE) version [v5.0], focusing specifically on radiation dermatitis grading (21).
  * Radiation dermatitis will be assessed weekly (Day 1,7,14,21,28,35) by the attending radiation oncologist throughout the course of treatment, with documentation in MOSAIQ (radiation oncology information system) of onset, peak severity, and any treatment-related complications or interruptions.
  * CTCAE grading will be used to classify skin reactions as follows:
  * Grade 1: Faint erythema or dry desquamation
  * Grade 2: Moderate to brisk erythema; patchy moist desquamation mostly in skin folds
  * Grade 3: Moist desquamation in non-skin-fold areas; bleeding with minor trauma
  * Grade 4: Skin necrosis or ulceration of full-thickness dermis
  * Grade 5: Death (extremely rare in this context)
Number of patients with maximum dermatitis grade during treatment. | Day 7, 14, 21, 28, 35 of radiotherapy
  Number of patients with maximum dermatitis grade during treatment.
Number of patients with incidence of moist desquamation. | Day 7, 14, 21, 28, 35 of radiotherapy treatment
  Incidence of moist desquamation will be assessed weekly by the attending radiation oncologist throughout the course of treatment, with documentation in MOSAIQ (radiation oncology information system)
Number of patients with treatment interruptions >3 days due to skin toxicity. | From beginning to end of radiotherapy treatment (Day 1 to Day 35)
  Any interruptions in radiotherapy treatment >3 days due to skin toxicity
Patient-reported outcomes from EORTC QLQ-HN35 for each participant | At baseline (Day 1), mid-treatment (Day 17) at end of radiotherapy treatment (Day 35).
  * The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) H&N35 is a questionnaire developed specifically for patients with head and neck cancer. It includes 35 questions grouped into 7 subscales covering pain, swallowing, senses (taste/smell), speech, social eating, social contact, and sexuality.
  * In addition, there are 10 individual items addressing issues such as dental problems, dry mouth, coughing, difficulty opening the mouth, sticky saliva, weight loss or gain, use of nutritional supplements, feeding tubes, and pain medication.
  * Interpretation of scores:
  Scores are from 1 to 4, where 1 reflects "not at all" and 4 is "very much". Higher scores on the functional and global health scales indicate better functioning and well-being, whereas higher scores on the symptom scales reflect greater symptom burden or difficulty.
Global health/quality of life impact (QLQ-C30) for every participant | At baseline (Day 1), mid-treatment (Day 17) at end of radiotherapy treatment (Day 35).
  • The European Organisation for Research and Treatment of Cancer (EORTC) QLQ C30. This questionnaire includes 30 items, that describe 5 functioning scales (physical, role, emotional, cognitive, and social functioning), 3 symptom scales (fatigue, nausea/vomiting, and pain), and 6 single items symptoms (dyspnoea, insomnia, loss of appetite, constipation, diarrhoea, and financial difficulties). Interpretation of scores. Scores are from 1 to 4, where 1 reflects "not at all" and 4 is "very much". Higher scores on the symptom scales reflect greater symptom burden or difficulty.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bjordal K, Hammerlid E, Ahlner-Elmqvist M, de Graeff A, Boysen M, Evensen JF, Biorklund A, de Leeuw JR, Fayers PM, Jannert M, Westin T, Kaasa S. Quality of life in head and neck cancer patients: validation of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-H&N35. J Clin Oncol. 1999 Mar;17(3):1008-19. doi: 10.1200/JCO.1999.17.3.1008. PMID 10071296
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Tayyib NA. Prophylactic Use of Mepitel(R) Film to Prevent Radiation-Induced Moist Desquamation in Cancer Patients. Cureus. 2023 Jul 20;15(7):e42186. doi: 10.7759/cureus.42186. eCollection 2023 Jul. PMID 37601988
- [Background] Wong HCY, Lee SF, Caini S, Chan AW, Kwan JYY, Waddle M, Sonis S, Herst P, Alcorn S, Bonomo P, Wong C, Corbin K, Choi JI, Rembielak A, AlKhaifi M, Marta GN, Rades D, van den Hurk C, Wolf JR, Chan RJ, Schmeel LC, Lock M, Hijal T, Cao J, Kim H, Chow E. Barrier films or dressings for the prevention of acute radiation dermatitis in breast cancer: a systematic review and network meta-analysis. Breast Cancer Res Treat. 2024 Oct;207(3):477-496. doi: 10.1007/s10549-024-07435-2. Epub 2024 Aug 7. PMID 39112742
- [Background] Yee C, Lam E, Gallant F, Karam I, Czarnota G, Soliman H, Wong G, Drost L, Vesprini D, Rakovitch E, Wronski M, Leung E, Szumacher E, Carothers K, Pon K, Gonzales G, Easton L, Lewis D, Zhang L, Chow E. A Feasibility Study of Mepitel Film for the Prevention of Breast Radiation Dermatitis in a Canadian Center. Pract Radiat Oncol. 2021 Jan-Feb;11(1):e36-e45. doi: 10.1016/j.prro.2020.09.004. Epub 2020 Sep 17. PMID 32949772
- [Background] Fernandez-Castro M, Martin-Gil B, Pena-Garcia I, Lopez-Vallecillo M, Garcia-Puig ME. Effectiveness of semi-permeable dressings to treat radiation-induced skin reactions. A systematic review. Eur J Cancer Care (Engl). 2017 Nov;26(6). doi: 10.1111/ecc.12685. Epub 2017 Apr 18. PMID 28417508
- [Background] Iacovelli NA, Torrente Y, Ciuffreda A, Guardamagna VA, Gentili M, Giacomelli L, Sacerdote P. Topical treatment of radiation-induced dermatitis: current issues and potential solutions. Drugs Context. 2020 Jun 12;9:2020-4-7. doi: 10.7573/dic.2020-4-7. eCollection 2020. PMID 32587626
- [Background] Tsai PC, Liu YC, Li TS, Hsu FT, Lee YH, Chiang IT, Chang Y, Lee CH. Clinical Effect of Moisturized Skin Care on Radiation Dermatitis of Head and Neck Cancer. In Vivo. 2023 Nov-Dec;37(6):2776-2785. doi: 10.21873/invivo.13389. PMID 37905662
- [Background] Zenda S, Ishi S, Kawashima M, Arahira S, Tahara M, Hayashi R, Kishimoto S, Ichihashi T. A Dermatitis Control Program (DeCoP) for head and neck cancer patients receiving radiotherapy: a prospective phase II study. Int J Clin Oncol. 2013 Apr;18(2):350-5. doi: 10.1007/s10147-012-0385-9. Epub 2012 Feb 15. PMID 22350025
- [Background] Zenda S, Ishi S, Akimoto T, Arahira S, Motegi A, Tahara M, Hayashi R, Asanuma C. DeCoP, a Dermatitis Control Program using a moderately absorbent surgical pad for head and neck cancer patients receiving radiotherapy: a retrospective analysis. Jpn J Clin Oncol. 2015 May;45(5):433-8. doi: 10.1093/jjco/hyv010. Epub 2015 Feb 11. PMID 25673153
- [Background] Agnihotri V, Kshirsagar AY. To assess the incidence of radiation dermatitis among the cancer patients receiving radiotherapy. Int J Nurs Med Invest. 2018;3(3):107-110.